CLINICAL TRIAL: NCT04692155
Title: Phase Ib/II Trial of Ublituximab and Umbralisib With CHOP (U2-CHOP) Followed by U2 Maintenance (U2-CHOP-U2) in Previously Untreated Mantle Cell Lymphoma (MCL)
Brief Title: Clinical Trial of Ublituximab and Umbralisib With CHOP (U2-CHOP) Followed by U2 Maintenance (U2-CHOP-U2) in Previously Untreated Mantle Cell Lymphoma (MCL)
Acronym: CHOP U2
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: FDA hold
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amitkumar Mehta, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300006404
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Mantle Cell Lymphoma
Keywords: Ublituximab; Umbralisib; TGR-1202; TG-1101
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ublituximab; umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- phase 1b and phase 2 (Experimental): for phase 1 B portion, Ublitixumab will be given IV at dosage 900mg from Cycle 1 Day1 till cycle 6. If investigator decides to continue the treatment as maintenance, Ublitixumab will be given IV every 8 weeks for 24 months Umbralisib (800mg) will be given orally once a day within 30 minutes of a meal from Cycle 1 Day1 till cycle 6.If investigator decides to continue the treatment as maintenance,• Umbralisib will be given at orally daily for 24 months.
  Chemotherapy combination of CHOP-cyclophosphamide IV 750mg/m2 for Age <70 years, 500 mg/m2 for Age>70 years doxorubicin IV 50mg/m2for Age <70 years, 25 mg/m2 for Age>70 years , and vincristine IV 1mg/m2 (max 2mg)) are administered on Cycle 1 day 1 till Cycle 6. Prednisone 50-100mg will be given orally on days 1 through 5 of every cycle.
  For Phase II portion- Once Umbralisib dose is defined in phase Ib, the study will expand to phase II portion after SMC/DSMB (Safety monitoring committee/Data Safety Monitoring Committee) agrees.
  Interventions: Drug: Ublituximab; Drug: Umbralisib

INTERVENTIONS:
Drug: Ublituximab — Ublituximab (900mg) will be administered as an intravenous infusion through a dedicated line.
  Other Names: TG-1101
Drug: Umbralisib — Umbralisib(800mg)will be administered orally once daily within 30 minutes of starting a meal.
  Other Names: TGR-1202

SUMMARY:
This is a single arm, multi-center, open label Phase Ib/II trial in adult patients with newly diagnosed Mantle Cell Lymphoma (MCL)(Stage II-IV). The Diagnosis of MCL (Stage II, III, IV) is supported by histology and over expression of cyclin D1 or by FISH (fluorescent in situ hybridization). In the proposed study, the primary endpoint is to estimate the biological response rate of the combination of Umbralisib at dose 800 mg with Ublituximab (900mg)-Cyclophosphamide, Doxorubicin, Vincristine and Prednisone (CHOP), but a phase Ib portion with dose de-escalation at two does level (800 and 600 mg) will be built in to further confirm its safety and tolerability. Treatment will be administered on an outpatient basis in 3-week (21 day) cycles. Once Umbralisib dose is defined in phase Ib, the study will expand to phase II portion after SMC/DSMB (Safety monitoring committee/Data Safety Monitoring Committee) agreement.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL) is an aggressive and incurable hematologic malignancy with incidence of MCL increases with age (average age is 68 years) and is more common in males. Majority of the patients presents with advanced systemic and symptomatic disease requiring aggressive chemotherapy. Although some patients with MCL can have indolent course, majority of them pursue an aggressive course. Most patients with MCL presents with non-bulky lymphadenopathy and advanced stage with frequent extra-nodal involvement. In general, MCL carries an aggressive course with very poor outcome. MCL has wide spectrum of clinical presentation ranging from indolent disease to symptomatic aggressive disease. The initial treatment of MCL depends on many disease and patient related factors. Advanced, biologically aggressive ( by histology markers) disease in a young and fit patient needs aggressive/intense induction, Autologus stem cell transplant (ASCT) consolidation and maintenance treatment. While unfit patient usually is offered less intense treatment followed by maintenance treatment.

Investigational drugs ublituximab & umbralisib are highly active in various B cell lymphomas. Umbralisib is a highly-specific and orally available dual inhibitor of phosphoinositide-3-kinase (PI3K) delta (δ) and casein kinase 1 epsilon (CK1ε) with nanomolar inhibitory potency, and high selectivity over the alpha, beta, and gamma Class I isoforms of PI3K. The PI3Ks are a family of enzymes involved in various cellular functions, including cell proliferation and survival, cell differentiation, intracellular trafficking and immunity. The delta isoform of PI3K is highly expressed in cells of hematopoietic origin, and strongly upregulated, and often mutated in various hematologic malignancies.

Ublituximab is a novel third generation chimeric anti-CD20 monoclonal antibody bioengineered for potent activity, exhibiting a unique glycosylation profile with a low fucose content, designed to induce superior antibody-dependent cytotoxicity (ADCC). Ublituximab exhibits competitive complement-dependent cytotoxicity (CDC), on par with rituximab, and has also been demonstrated to induce programmed cell death (PCD) upon binding to the CD20 antigen on B-lymphocytes.

Pre-Clinical Development Of Ublituximab:

The antitumor effect of ublituximab was compared to that of rituximab with chemotherapy in follicular lymphoma (FL), and mantle cell lymphoma (MCL) xenograft murine models. Single agent ublituximab demonstrated dose-related anti-tumor activity with 100% tumor growth inhibition in the FL xenograft at a dose of 100mg/kg, and a superior tumor growth delay (21 days) compared to rituximab. Ublituximab also demonstrated superior anti-tumor activity compared to rituximab against MCL xenografts at all dose levels (Esteves IT, 2011).

Ublituximab in Combination with Umbralisib :

The combination of Ublituximab and Umbralisib is being evaluated in various clinical trials. The preliminary data suggests that the combination is safe and well tolerated. Results of a Phase I/Ib study of the combination of ublituximab + umbralisib (U2) in patients with relapsed or refractory Non-Hodgkin Lymphoma(NHL) and Chronic lymphocytic Leukemia(CLL) have been reported. Overall, results from this study suggest that the U2 regimen is well tolerated and active in patients with relapsed or refractory hematologic malignancies.

Rationale for this Study:

This is a Single arm, multi-center, open label Phase II trial with safety lead in Adult patients with newly diagnosed Mantle Cell Lymphoma (MCL)(Stage II-IV). MCL majority, is an aggressive and incurable lymphoma. As it is the lymphoma of elderly, aggressive treatment approaches like aggressive induction treatments and ASCT may be more risky in this population. Majority of these patients are treated with less intense approach like Rituximab-Bendamustine (BR), R-CHOP or VR-CAP. Nearly all the patients are treated with Rituximab maintenance after these induction approaches.

In this study, we will explore combination of novel CD20 monoclonal antibody (Ublituximab) with CHOP and a novel highly active PI3K inhibitor (Umbralisib) in ASCT ineligible untreated advanced MCL. Umbralisib is highly active in various B cell lymphomas. The combination of Ublituximab and Umbralisib is being evaluated in two signature clinical trials. The preliminary data suggests that the combination is safe and well tolerated. To improve upon the back bone of R-CHOP, we want to explore U2-CHOP (Ublituximab with Umbralixib)-CHOP followed by U2 maintenance in ASCT in eligible patients. Both the study agents (U2) are highly active in lymphomas. Study hypothesis is to improve rates of complete response at the end of induction treatment with this novel combination.

Study Objectives:

* To determine the safety of Umbralisib and Ublituximab in combination with CHOP chemotherapy for newly diagnosed MCL.
* To determine the efficacy of U2-CHOP in terms of Complete Response rates (CRR) in patients with untreated MCL after induction phase (6 cycles of U2-CHOP) by PET/CT response assessment criteria by Cheson 2014.
* To characterize the toxicity profile of U2-CHOP induction followed by U2 maintenance in newly diagnosed Mantle Cell Lymphoma (MCL) patients.
* To determine rates of Overall response rate, disease control rate
* Overall survival and progression free survival
* To explore minimal residual disease (MRD) negative rates at the end of induction treatment

ELIGIBILITY:
Inclusion Criteria:

* Males or female patients >18 years of age
* Diagnosis of MCL (Ann Arbor Stage II, III, IV) as supported by histology and over expression of cyclin D1 (in association with CD20 and CD5) or evidence of t(11;14) by FISH (fluorescent in situ hybridization) with indication of initiation of therapy.
* At least one LN of >1.5 cm size as index/measurable site of disease
* No prior anti-cancer therapy for MCL
* Not eligible for bone marrow transplantation/ASCT (assessed by treating physician due to comorbidities) or not interested in bone marrow transplant/ASCT (clear documentation of patient's unwillingness to pursue transplant)
* Eastern cooperative Oncology Group (ECOG) performance status: 0,1 or 2
* Absolute neutrophil count (ANC) >1500/microL (>1000 if bone marrow involvement with MCL) within 28 days prior to initiation of therapy. Growth factors are not permitted for the purpose of meeting eligibility criteria.
* Platelets >100000 cells/uL (>75000 cells/uL if bone marrow involvement with MCL) within 28 days prior to initiation of therapy. Growth factors are not permitted for the purpose of meeting eligibility criteria.
* Hemoglobin >9.0 gm/dL (>8.0 gm/dL if bone marrow involvement with MCL) within 28 days prior to initiation of therapy. Growth factors are not permitted for the purpose of meeting eligibility criteria.
* Alanine transaminase (ALT)/Aspartate Transaminase (AST) <2.5 X Upper limit of Normal (ULN) if no liver involvement or ≤ 5 x the ULN if known liver involvement within 28 days prior to initiation of therapy
* Total Bilirubin <1.5X ULN within 28 days prior to initiation of therapy (Except in Gilbert's disase <3XULN is allowed)
* Calculated Creatinine Clearance >35 mL/min by Cockcroft-Gault Equation
* Male patients must agree to use an acceptable method of contraception for the entire duration of study and for 4 months after the last dose of either study drug.
* All patients (or their legal representative) must have signed an informed consent indicating that they are willing to participate in the study and are willing to follow the procedure required by the study in accordance with federal, local and institutional guidelines.
* Female patients who are not of child-bearing potential, and female patients of child-bearing potential who have a negative serum pregnancy test within 3 days prior to initial trial treatment Female patients of child-bearing potential and all male partners must consent to use a medically acceptable method of contraception throughout the study period and for 4 months after the last dose of either study drug.

Exclusion Criteria:

* Any prior anti-neoplastic therapy for MCL
* CNS involvement by MCL
* Malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, non-melanomatous skin cancer or localized thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection/radiation or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.
* If patient has received prior anthracycline therapy, the cumulative anthracycline dose should be <150mg/m2 of doxorubicin equivalent
* H/O prior Allogeneic transplantation or autologous stem cell transplantation for any other reason.
* Use of immunosuppressive therapy (e.g. cyclosporine A, tacrolimus or high dose steroids). Patients receiving steroids must be at a dose of <10mg/day prednisone (or equivalent) within 7 days of the first day of the study treatment administration. Patients are allowed to use topical or inhaled corticosteroids.
* Concurrent any systemic anticancer therapy for any other cancer (chemotherapy, radiation, surgery, immunotherapy, biologic therapy, hormonal therapy, investigational therapy or tumor embolization).
* Uncontrolled Diabetes Mellitus, Hyperglycemia (patients with endocrine consultation and proper plan with reasonable control of blood sugars are allowed)
* Any uncontrolled auto-immune condition like hepatitis, colitis, pneumonitis etc which in view of investigator is high risk to be treated on this combination
* History of stroke or intracranial hemorrhage within 6 months of the date of study treatment administration (unless complete and full recovery)
* Chronic or current active infections requiring intravenous antibiotics, antifungal or antiviral treatment or exposure to live vaccines within 30 days of study treatment.
* Known HIV infection or history of HIV.
* Evidence of Hepatitis B or Hepatitis C infection or risk of reactivation. HBV DNA or HCV RNA evidence of chronic active Hepatitis B (HBV, not including patients with prior hepatitis B vaccination; or positive serum Hepatitis B antibody) or chronic active Hepatitis C infection (HCV), active cytomegalovirus (CMV), or known history of HIV. If HBc antibody is positive, the subject must be evaluated for the presence of HBV DNA by PCR. If CMV IgG or IgM is reactive, the subject must be evaluated for the presence of CMV DNA by PCR. If HCV antibody is positive, the subject must be evaluated for the presence of HCV RNA by PCR. See Appendix: HEPATITIS B SEROLOGIC TEST RESULTS. Subjects with positive HBc antibody and negative HBV DNA by PCR are eligible. Subjects with positive HCV antibody and negative HCV RNA by PCR are eligible. Subjects who are CMV IgG or CMV IgM positive but who are CMV DNA negative by PCR are eligible.
* Known history of drug-induced liver injury, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by stones, cirrhosis of the liver
* Any severe and/or uncontrolled medical conditions or other conditions that could affect participation in the study such as:
* Symptomatic, or history of documented congestive heart failure (New York Heart Association functional classification II-IV)[see Appendix: NYHA Classifications]
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, CHF, or myocardial infarction within 6 months of enrollment.
* Concomitant use of medication known to cause QT prolongation or torsades de pointes should be used with caution and at investigator discretion.
* Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), angioplasty, cardiac or vascular stenting within 6 months of enrollment.
* Cardiac ejection fraction (EF) <45%.
* Current NY heart association Class II to IV congestive heart failure or uncontrolled arrhythmia
* Presence of an abnormal ECG that is clinically meaningful. Patients with QTc interval >450 for males and >470 milliseconds for females are excluded (corrected by Fridericia).
* Currently pregnant or breast feeding.
* Unable to swallow and retain oral medication, malabsorption syndrome, disease significantly affecting GI function, total resection of stomach or small bowel, ulcerative colitis, symptomatic IBD or complete or partial obstruction.
* Anaphylaxis, excluding infusion related reactions, to monoclonal antibody/Rituximab in past.
* Any condition that would, in investigator's judgment, interfere with full participation in the study, including administration of study medication/chemotherapy, attending study visits, pose a risk to the patient or interfere with interpretation of study data.
* Inability to comprehend or unwilling to sign the ICF.
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 21 days prior to registration
* Contraindication or intolerance to required supportive care medications (pegfilgrastim, acyclovir or bactrim/dapsone/pentamidine/atovaquone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amitkumar Mehta, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b and Phase 2: for phase 1 B portion, Ublitixumab will be given IV at dosage 900mg from Cycle 1 Day1 till cycle 6. If investigator decides to continue the treatment as maintenance, Ublitixumab will be given IV every 8 weeks for 24 months Umbralisib (800mg) will be given orally once a day within 30 minutes of a meal from Cycle 1 Day1 till cycle 6.If investigator decides to continue the treatment as maintenance,• Umbralisib will be given at orally daily for 24 months.
  Chemotherapy combination of CHOP-cyclophosphamide IV 750mg/m2 for Age <70 years, 500 mg/m2 for Age>70 years doxorubicin IV 50mg/m2for Age <70 years, 25 mg/m2 for Age>70 years , and vincristine IV 1mg/m2 (max 2mg)) are administered on Cycle 1 day 1 till Cycle 6. Prednisone 50-100mg will be given orally on days 1 through 5 of every cycle.
  For Phase II portion- Once Umbralisib dose is defined in phase Ib, the study will expand to phase II portion after SMC/DSMB (Safety monitoring committee/Data Safety Monitoring Committee) agrees.
  Ublituximab: Ublituximab (900mg) will be administered as an intravenous infusion through a dedicated line.
  Umbralisib: Umbralisib(800mg)will be administered orally once daily within 30 minutes of starting a meal.
Period: Overall Study
Arm/Group | Phase 1b and Phase 2
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Phase 1b and Phase 2
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Remission at the End of Induction Treatment
Description: In the proposed study, the primary endpoint is to estimate the biological response rate of the combination of Umbralisib at dose 800 mg with Ublituximab (900mg)-CHOP, but a phase Ib portion with dose de-escalation at two does level (800 and 600 mg) will be built in to further confirm its safety and tolerability. Rate of complete remission at the end of induction treatment (U2-CHOP X 6 cycles) per PET/CT assessment criteria for Lymphoma (Cheson et al, 2014).Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 10 months
Population: The patient died because of COVID infection. Not related to the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b and Phase 2
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: To determine the efficacy of U2-CHOP in terms of PFS in patients with untreated MCL after induction phase (6 cycles of U2-CHOP) by PET/CT response assessment criteria by Cheson 2014
Time Frame: Baseline through 3 years
Population: The patient died because of COVID infection. Not related to the study drug. No data was collected.
Arm/Group | Phase 1b and Phase 2
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (OS)
Description: To determine the efficacy of U2-CHOP in terms of OS in patients with untreated MCL after induction phase (6 cycles of U2-CHOP) by PET/CT response assessment criteria by Cheson 2014
Time Frame: Baseline through 3 years
Population: The patient died because of COVID infection. Not related to the study drug. No data was collected
Arm/Group | Phase 1b and Phase 2
Number analyzed (Participants) | 0

4. Secondary Outcome: Rate of Overall Response Rate (Complete Response CR+ Partial Response PR)
Description: To determine the efficacy of U2-CHOP in terms of Overall Response rates (ORR) in patients with untreated MCL after induction phase (6 cycles of U2-CHOP) by PET/CT response assessment criteria by Cheson 2014.
Time Frame: Baseline through 3 years
Population: The patient died because of COVID infection. Not related to the study drug. No data was collected
Arm/Group | Phase 1b and Phase 2
Number analyzed (Participants) | 0

5. Secondary Outcome: Rate of Disease Control Rate (CR+PR+SD)
Description: To determine the efficacy of U2-CHOP in terms of Rate of disease control rate in patients with untreated MCL after induction phase (6 cycles of U2-CHOP) by PET/CT response assessment criteria by Cheson 2014
Time Frame: Baseline through 3 years
Population: The patient died because of COVID infection. Not related to the study drug. No data was collected
Arm/Group | Phase 1b and Phase 2
Number analyzed (Participants) | 0

6. Secondary Outcome: Rate of Minimal Residual Disease MRD Negativity at the End of Induction Treatment
Description: MRD status is a future exploratory endpoint for this trial. Peripheral blood samples are required at the end of induction treatment
Time Frame: Baseline through 2 years
Population: The patient died because of COVID infection. Not related to the study drug. No data was collected
Arm/Group | Phase 1b and Phase 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Phase 1b and Phase 2
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT04692155/Prot_SAP_002.pdf